CLINICAL TRIAL: NCT04223232
Title: An Open-Label, Single-Dose, Single-Period Study Designed to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]-MD1003 in Healthy Male Subjects
Brief Title: Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]-MD1003 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedDay Pharmaceuticals SA (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MD1003CT2019-03MB
Record Dates: First submitted 2019-12-13; First posted 2020-01-10 (Actual); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MD1003 (Experimental): radiolabeled 14C MD1003 (High Dose Biotin) 100mg
  Interventions: Drug: [14C]-MD1003

INTERVENTIONS:
Drug: [14C]-MD1003 — single oral dose of 100mg [14C]-MD1003

SUMMARY:
This single-center, open-label, non randomized Phase I study is being conducted to investigate the pharmacokinetics, mass balance and metabolite profiling and identification after a single oral dose of 100mg of [14C]-MD1003 in 6 healthy males subjects. The radioactivity will be followed in the blood, urine and faeces to study MD1003 metabolism.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males
2. Age 30 to 65 years of age at the time of signing informed consent
3. Body mass index (BMI) of 18.0 to 30.0 kg/m2 as measured at screening
4. Must be willing and able to communicate and participate in the whole study
5. Must have regular bowel movements (ie average stool production of ≥1 and ≤3 stools per day)
6. Must provide written informed consent
7. Must agree to adhere to the contraception requirements of the protocol

Exclusion Criteria:

1. Subjects who have received any IMP in a clinical research study within the 90 days prior to Day 1
2. Subjects who are study site employees, or immediate family members of a study site or sponsor employee
3. Subjects who have previously been enrolled in this study
4. History of any drug or alcohol abuse in the past 2 years
5. Regular alcohol consumption in males >21 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 Units = 125 mL glass of wine, depending on type)
6. A confirmed positive alcohol breath test at screening or admission
7. Current smokers and those who have smoked within the last 12 months. A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission
8. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
9. Subjects with pregnant or lactating partners
10. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic X-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, shall participate in the study
11. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator or delegate at screening
12. Clinically significant abnormal clinical chemistry, haematology or urinalysis as judged by the investigator. Subjects with Gilbert's Syndrome are allowed
13. Confirmed positive drugs of abuse test result (drugs of abuse tests are listed in the protocol)
14. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
15. Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance of <80 mL/min using the Cockcroft-Gault equation
16. History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder, as judged by the investigator
17. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
18. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active
19. Donation or loss of greater than 400 mL of blood within the previous 3 months
20. Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than 4 g of paracetamol per day), herbal remedies, vitamin B5 or dietary supplements containing lipoic acid in the 14 days before IMP administration. Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as determined by the PI
21. Subjects who have had any intake of biotin (including as a nutritional supplement) in the 14 days before IMP administration
22. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Somasekhara Menakuru, MS, MRCS, Principal Investigator — Quotient Sciences Nottingham, UK, NG116JS
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MD1003
Started | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | MD1003
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6

OUTCOME MEASURES:

1. Primary Outcome: Mass Balance Recovery of Total Radioactivity: CumAe (Urine)
Description: Cumulative amount of total radioactivity excreted in urine Measured at 0/12/24/48/72/96/120/144/168/192/216/240/264/288/312 hours
Time Frame: Pre-dose to 312 hours post-dose
Measure: Mean (Standard Deviation); unit: mg equiv
Arm/Group | MD1003
Number analyzed (Participants) | 6
mg equiv | 70.9 (16.9)

2. Primary Outcome: Mass Balance Recovery of Total Radioactivity: Cum%Ae (Urine)
Description: Cumulative amount of total radioactivity excreted in urine expressed as a percentage of the radioactive dose administered Measured at 0/0.5/1/1.5/2/3/4/6/8/12/18/24/36/48/72/96/120/144/168/192/216/240/264/288/312 hours.
Time Frame: Pre-dose to 312 hours post dose
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | MD1003
Number analyzed (Participants) | 6
percentage | 70.786 (16.874)

3. Primary Outcome: Mass Balance Recovery of Total Radioactivity: CumAe (Faeces)
Description: Cumulative amount of total radioactivity excreted in faeces Measured at 0/0.5/1/1.5/2/3/4/6/8/12/18/24/36/48/72/96/120/144/168/192/216/240/264/288/312 hours.
Time Frame: Pre-dose to 312 hours post-dose
Measure: Mean (Standard Deviation); unit: mg equiv
Arm/Group | MD1003
Number analyzed (Participants) | 6
mg equiv | 16.0 (8.63)

4. Primary Outcome: Mass Balance Recovery of Total Radioactivity: Cum%Ae (Faeces)
Description: Cumulative amount of total radioactivity excreted in faeces expressed as a percentage of the radioactive dose administered Measured at 0/0.5/1/1.5/2/3/4/6/8/12/18/24/36/48/72/96/120/144/168/192/216/240/264/288/312 hours.
Time Frame: Pre-dose to 312 hours post dose
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | MD1003
Number analyzed (Participants) | 6
percentage | 16.009 (8.617)

5. Primary Outcome: Mass Balance Recovery of Total Radioactivity: CumAe(Total)
Description: Cumulative amount of total radioactivity excreted in urine and faeces combined Measured at 0/0.5/1/1.5/2/3/4/6/8/12/18/24/36/48/72/96/120/144/168/192/216/240/264/288/312 hours.
Time Frame: Pre-dose to 312 hours post dose
Measure: Mean (Standard Deviation); unit: mg equiv
Arm/Group | MD1003
Number analyzed (Participants) | 6
mg equiv | 86.9 (9.25)

6. Primary Outcome: Mass Balance Recovery of Total Radioactivity: Cum%Ae (Total)
Description: Cumulative amount of total radioactivity excreted in urine and faeces combined expressed as a percentage of the radioactive dose administered Measured at 0/0.5/1/1.5/2/3/4/6/8/12/18/24/36/48/72/96/120/144/168/192/216/240/264/288/312 hours.
Time Frame: Pre-dose to 312 hours post dose
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | MD1003
Number analyzed (Participants) | 6
percentage | 86.795 (9.235)

7. Secondary Outcome: Time Prior to the First Measurable Concentration (Tlag) for MD1003, Bisnorbiotin, Biotin Sulfoxide and Total Radioactivity
Description: Measured at 0/1/1.5/2/3/4/6/8/12/18/24/36/48/72/96/120/144/168 hours.
Time Frame: Pre-dose to 168 hours
Measure: Mean (Full Range); unit: hours
Arm/Group | MD1003
Number analyzed (Participants) | 6
hours
  MD1003 | 0.083 [0.00 to 0.50]
  Bisnorbiotin | 0.753 [0.50 to 1.50]
  Biotin Sulfoxide | 0.753 [0.50 to 1.50]
  Total radioactivity | 0.000 [0.00 to 0.00]

8. Secondary Outcome: Time of Maximum Plasma Concentration (Tmax) for MD1003, Bisnorbiotin, Biotin Sulfoxide and Total Radioactivity
Description: Measured at 0/1/1.5/2/3/4/6/8/12/18/24/36/48/72/96/120/144/168 hours.
Time Frame: Pre-dose to 168 hours
Measure: Mean (Full Range); unit: hours
Arm/Group | MD1003
Number analyzed (Participants) | 6
hours
  MD1003 | 2.086 [1.52 to 3.00]
  Bisnorbiotin | 4.011 [3.00 to 6.00]
  Biotin Sulfoxide | 2.667 [2.00 to 4.00]
  Total radioactivity | 2.667 [2.00 to 4.00]

9. Secondary Outcome: Maximum Plasma Concentration (Cmax) for MD1003, Bisnorbiotin, Biotin Sulfoxide and Total Radioactivity
Description: Measured at 0/1/1.5/2/3/4/6/8/12/18/24/36/48/72/96/120/144/168 hours.
Time Frame: Pre-dose to 168 hours
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | MD1003
Number analyzed (Participants) | 6
ng/mL
  MD1003 | 387 [325 to 416]
  Bisnorbiotin | 45.5 [26.4 to 59.0]
  Biotin Sulfoxide | 14.5 [9.70 to 18.9]
  Total radioactivity | 501 [469 to 543]

10. Secondary Outcome: Area Under Plasma Concentration Curve From 0 Time to Last Measurable Concentration (AUC(0-last)) for MD1003, Bisnorbiotin, Biotin Sulfoxide and Total Radioactivity
Description: Measured at 0/1/1.5/2/3/4/6/8/12/18/24/36/48/72/96/120/144/168 hours.
Time Frame: Pre-dose to 168 hours
Measure: Mean (Full Range); unit: ng.h/mL
Arm/Group | MD1003
Number analyzed (Participants) | 6
ng.h/mL
  MD1003 | 3350 [2750 to 4480]
  Bisnorbiotin | 514 [246 to 890]
  Biotin Sulfoxide | 74.3 [47.4 to 123]
  Total radioactivity | 2690 [2490 to 3310]

11. Secondary Outcome: Area Under Plasma Concentration Curve From 0 Time Extrapolated to Infinity (AUC(0-inf)) for MD1003 and Total Radioactivity
Description: Measured at 0/1/1.5/2/3/4/6/8/12/18/24/36/48/72/96/120/144/168 hours.
Time Frame: Pre-dose to 168 hours
Population: For total radioactivity: for 3 patients, extrapolated portion of AUC(0-inf) >20%.
Measure: Mean (Full Range); unit: ng.h/mL
Arm/Group | MD1003
Number analyzed (Participants) | 6
ng.h/mL
  MD1003 | 3650 [3010 to 4750]
  Total radioactivity: number analyzed (Participants) | 3
  Total radioactivity | 2850 [2670 to 3060]

12. Secondary Outcome: Percentage of AUC(0-extrap) Extrapolated Beyond the Last Measurable Concentration for MD1003 and Total Radioactivity
Description: Measured at 0/1/1.5/2/3/4/6/8/12/18/24/36/48/72/96/120/144/168 hours.
Time Frame: Pre-dose to 168 hours
Population: For total radioactivity: for 3 patients, extrapolated portion of AUC(0-inf) >20%.
Measure: Mean (Full Range); unit: percentage of AUC(0-extrap)
Arm/Group | MD1003
Number analyzed (Participants) | 6
percentage of AUC(0-extrap)
  MD1003 | 8.405 [5.76 to 11.33]
  Total radioactivity: number analyzed (Participants) | 3
  Total radioactivity | 15.171 [10.15 to 18.82]

13. Secondary Outcome: Area Under Plasma Concentration Curve From 0 Time to Last Measurable Concentration (AUC(0-12)) for MD1003, Bisnorbiotin, Biotin Sulfoxide and Total Radioactivity
Description: Measured at 0/1/1.5/2/3/4/6/8/12/18/24/36/48/72/96/120/144/168 hours.
Time Frame: Pre-dose to 168 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | MD1003
Number analyzed (Participants) | 6
ng.h/mL
  MD1003 | 1760 (16.50)
  Bisnorbiotin | 279 (26.4)
  Biotin Sulfoxide | 90.1 (23.7)
  Total radioactivity | 2680 (10.6)

14. Secondary Outcome: Lambda-z for MD1003, Bisnorbiotin, Biotin Sulfoxide and Total Radioactivity
Description: Measured at 0/1/1.5/2/3/4/6/8/12/18/24/36/48/72/96/120/144/168 hours.
Time Frame: Pre-dose to 168 hours
Measure: Mean (Full Range); unit: 1/Hours
Arm/Group | MD1003
Number analyzed (Participants) | 6
1/Hours
  MD1003 | 0.02302 [0.0180 to 0.0269]
  Bisnorbiotin | 0.02251 [0.0165 to 0.0285]
  Biotin Sulfoxide | 0.11829 [0.0324 to 0.1683]
  Total radioactivity | 0.20071 [0.0756 to 0.3762]

15. Secondary Outcome: Plasma Clearance (CL/F) for MD1003
Description: Measured at 0/1/1.5/2/3/4/6/8/12/18/24/36/48/72/96/120/144/168 hours.
Time Frame: Pre-dose to 168 hours
Measure: Mean (Full Range); unit: mL/min
Arm/Group | MD1003
Number analyzed (Participants) | 6
mL/min | 465 [351 to 554]

16. Secondary Outcome: Plasma Clearance (Vz/F) for MD1003
Description: Measured at 0/1/1.5/2/3/4/6/8/12/18/24/36/48/72/96/120/144/168 hours.
Time Frame: Pre-dose to 168 hours
Measure: Mean (Full Range); unit: L
Arm/Group | MD1003
Number analyzed (Participants) | 6
L | 1230 [816 to 1560]

17. Secondary Outcome: Elimination Half Life (t1/2) for MD1003, Bisnorbiotin, Biotin Sulfoxide and Total Radioactivity
Description: Measured at 0//1/1.5/2/3/4/6/8/12/18/24/36/48/72/96/120/144/168 hours.
Time Frame: Pre-dose to 168 hours
Population: For Bisnorbiotin: terminal slopes could not be reliably determined for all, due to an unacceptable coefficient of determination (ie, R2 < 0.9).
  For Biotin sulfoxide: terminal slopes could not be reliably determined all, due to an unacceptable coefficient of determination (ie, R2 < 0.9) or insufficient data points after Cmax.
Measure: Mean (Full Range); unit: hours
Arm/Group | MD1003
Number analyzed (Participants) | 6
hours
  MD1003 | 30.625 [25.74 to 38.51]
  Bisnorbiotin: number analyzed (Participants) | 2
  Bisnorbiotin | 33.176 [24.29 to 42.065]
  Biotin Sulfoxide: number analyzed (Participants) | 3
  Biotin Sulfoxide | 10.010 [4.12 to 21.42]
  Total radioactivity | 4.502 [1.84 to 9.17]

18. Secondary Outcome: MPR Cmax for Bisnorbiotin and Biotin Sulfoxide
Description: MPR = metabolite to parent ratio Measured at 0/1/1.5/2/3/4/6/8/12/18/24/36/48/72/96/120/144/168 hours.
Time Frame: Pre-dose to 168 hours
Measure: Mean (Full Range); unit: none (ratio)
Arm/Group | MD1003
Number analyzed (Participants) | 6
none (ratio)
  Bisnorbiotin | 0.1327 [0.074 to 0.174]
  Biotin Sulfoxide | 0.0349 [0.028 to 0.044]

19. Secondary Outcome: MPR AUC(0-inf) for Bisnorbiotin and Biotin Sulfoxide
Description: MPR = metabolite to parent ratio Measured at 0/1/1.5/2/3/4/6/8/12/18/24/36/48/72/96/120/144/168 hours.
Time Frame: Pre-dose to 168 hours
Measure: Mean (Full Range); unit: none (ratio)
Arm/Group | MD1003
Number analyzed (Participants) | 6
none (ratio)
  Bisnorbiotin | 0.1731 [0.082 to 0.267]
  Biotin sulfoxide | 0.0204 [0.014 to 0.026]

20. Secondary Outcome: Whole Blood: Plasma Concentration Ratios of Total Radioactivity
Description: Total radioactivity in whole blood versus total radioactivity in plasma concentration ratios at time intervals following a single oral administration of 100mg [14C]-MD1003 Measured at 0/1/1.5/2/3/4/6/8/12/18/24/36/48/72/96/120/144/168 hours.
Time Frame: Pre-dose to 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: % radioactivity whole blood/plasma
Arm/Group | MD1003
Number analyzed (Participants) | 6
% radioactivity whole blood/plasma
  1 H | 1.298 (5.0)
  4 H | 0.931 (14.6)
  8 H | 1.365 (7.0)
  12 H | 1.708 (9.3)

21. Secondary Outcome: Number of Subjects With Adverse Events (AEs)
Description: 2 months
Time Frame: Overall period
Measure: Count of Participants; unit: Participants
Arm/Group | MD1003
Number analyzed (Participants) | 6
Participants | 2

22. Secondary Outcome: Number of Subjects With Adverse Drug Reactions as Assessed by Investigator
Time Frame: Overall period
Measure: Count of Participants; unit: Participants
Arm/Group | MD1003
Number analyzed (Participants) | 6
Participants | 0

23. Secondary Outcome: Change From Baseline in Systolic Blood Pressure in mmHg
Description: Change from baseline measure (defined as Day 1, pre-dose). Measured at screening/Pre-dose/1/4/24/72/168 hours.
Time Frame: Pre-dose to Day 10
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MD1003
Number analyzed (Participants) | 6
mmHg
  1H | 0.7 (4.9)
  4H | -3.5 (8.0)
  24H | -1.0 (10.3)
  72H | -2.8 (11.4)
  Discharge | 0.5 (6.9)

24. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure in mmHg
Description: Change from baseline measure (defined as Day 1, pre-dose). Measured at screening/Pre-dose/1/4/24/72/168 hours.
Time Frame: Pre-dose to Day 10
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MD1003
Number analyzed (Participants) | 6
mmHg
  1H | 3.2 (5.9)
  4H | 2.5 (6.1)
  24H | 2.0 (6.6)
  72H | -0.5 (5.8)
  Discharge | 4.7 (6.9)

25. Secondary Outcome: Change From Baseline in Heart Rate in Beats Per Minute
Description: Change from baseline measure (defined as Day 1, pre-dose). Measured at screening/Pre-dose/1/4/24/72/168 hours.
Time Frame: Pre-dose to Day 10
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | MD1003
Number analyzed (Participants) | 6
bpm
  1H | -3.7 (3.0)
  4H | -4.0 (4.8)
  24H | -2.5 (5.5)
  72H | -2.0 (6.0)
  Discharge | 3.3 (9.9)

26. Secondary Outcome: Change From Baseline in ECG (Electrocardiogram) QTcF Interval in Milliseconds
Description: Change from baseline measure (defined as Day 1, pre-dose). Measured at screening/Pre-dose/1/4/24/72/168 hours.
Time Frame: Pre-dose to Day 10
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | MD1003
Number analyzed (Participants) | 6
msec
  1H | 2.2 (6.9)
  4H | 2.7 (3.9)
  24H | 1.0 (4.6)
  Discharge | 1.0 (11.5)

ADVERSE EVENTS:
Time Frame: From Day -28 to Day 8
Arm/Group | MD1003
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MD1003 (N=6)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-09-12): https://cdn.clinicaltrials.gov/large-docs/32/NCT04223232/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/32/NCT04223232/SAP_001.pdf